CLINICAL TRIAL: NCT03268954
Title: A Phase 3, Randomized, Controlled, Open-label, Clinical Study of Pevonedistat Plus Azacitidine Versus Single-Agent Azacitidine as First-Line Treatment for Patients With Higher-Risk Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia, or Low-Blast Acute Myelogenous Leukemia
Brief Title: Pevonedistat Plus Azacitidine Versus Single-Agent Azacitidine as First-Line Treatment for Participants With Higher-Risk Myelodysplastic Syndromes (HR MDS), Chronic Myelomonocytic Leukemia (CMML), or Low-Blast Acute Myelogenous Leukemia (AML)
Acronym: PANTHER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pevonedistat-3001; 2017-000318-40 (EudraCT Number); U1111-1189-8055 (Other: World Health Organization); MOH_2018-02-04_002154 (Other: CRS); JapicCTI-183848 (Registry Identifier: JapicCTI); NCI-2017-02059 (Other: National Cancer Institute)
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndrome; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute
Keywords: Drug therapy
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Azacitidine; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azacitidine 75 mg/m^2 (Experimental): Participants were administered azacitidine 75 milligram per square meter (mg/m^2) intravenous (IV) or subcutaneous (SC) injection on Days 1 to 5, Days 8 and 9, in 28-day treatment cycles until disease progression or unacceptable toxicity or up to a maximum of 63 cycles.
  Interventions: Drug: Azacitidine
- Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 (Experimental): Participants were administered azacitidine 75 mg/m^2 IV or SC injection on Days 1 to 5, Days 8 and 9 and pevonedistat 20 mg/m^2 IV infusion, on Days 1, 3, and 5 in 28-day treatment cycles until disease progression or unacceptable toxicity or up to a maximum of 63 cycles.
  Interventions: Drug: Azacitidine; Drug: Pevonedistat

INTERVENTIONS:
Drug: Azacitidine — Azacitidine intravenous or subcutaneous formulation.
Drug: Pevonedistat — Pevonedistat intravenous infusion.
  Arms: Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2

SUMMARY:
The purpose of this study is to determine whether the combination of pevonedistat and azacitidine improves event-free survival (EFS) when compared with single-agent azacitidine. (An event is defined as death or transformation to AML in participants with MDS or CMML, whichever occurs first, and is defined as death in participants with low-blast AML).

DETAILED DESCRIPTION:
The drug being tested in this study is called pevonedistat. Pevonedistat is being tested to treat people with higher-risk myelodysplastic syndromes (HR MDS), chronic myelomonocytic leukemia (CMML) and low-blast acute myelogenous leukemia (AML) as a combination treatment with azacitidine. This study will look at the overall survival, event-free survival and response to treatment in people who take pevonedistat and azacitidine when compared to people who take single-agent azacitidine.

The study will enroll approximately 450 participants. Once enrolled, participants will be randomly assigned in 1:1 ratio (by chance, like flipping a coin) to one of the two treatment groups in 28-day treatment cycles:

* Pevonedistat 20 mg/m^2 and azacitidine 75 mg/m^2 combination
* Single-agent azacitidine 75 mg/m^2

All participants will receive azacitidine via intravenous or subcutaneous route. Participants randomized to the combination arm will also receive pevonedistat intravenous infusion.

This multi-center trial will be conducted Spain, Belgium, Brazil, Canada, Czech Republic, France, Germany, Israel, Italy, the United States, Australia, Greece, Japan, Mexico, Poland, Russia, Korea, Turkey, China and United Kingdom. The overall time to participate in this study is approximately 63 months. Participants will attend the end-of-treatment visit 30 days after the last dose of study drug or before the start of subsequent anti-neoplastic therapy if that occurs sooner.

Participants with HR MDS or CMML will have EFS follow-up study visits every month if their disease has not transformed to AML and they have not started subsequent therapy. Participants with low-blast AML will have response follow-up study visits every month until they relapse from CR or meet the criteria for PD. All participants will enter OS follow-up (contacted every 3 months) when they have confirmed transformation to AML (for participants with HR MDS or CMML at enrollment) or experienced PD (for participants with low-blast AML at study enrollment).

ELIGIBILITY:
Inclusion Criteria:

1. Has morphologically confirmed diagnosis of myelodysplastic syndromes (MDS) or CMML (i.e., with white blood cell [WBC] <13,000/microliter [mcL]) or low-blast acute myelogenous leukemia (AML).
2. Has MDS or CMML and must also have one of the following Prognostic Risk Categories, based on the Revised International Prognostic Scoring System (IPSS-R):

   * Very high (>6 points).
   * High (>4.5-6 points).
   * Intermediate (>3-4.5 points): a participant determined to be in the Intermediate Prognostic Risk Category is only allowable in the setting of >=5% bone marrow myeloblasts.
3. Eastern Cooperative Oncology Group (ECOG) status of 0, 1, or 2.
4. Participants with AML (20%-30% blasts) must have a treatment-related mortality (TRM) score >=4 for intensive, induction chemotherapy as calculated using the simplified model described by Walter and coworkers.

Calculation of TRM score:

* 0 for (age <61 years), +2 for (age 61-70 years), +4 for (age >=71 years).
* + 0 for (PS=0), +2 for (PS=1), +4 for (PS >1).
* + 0 for (platelets <50), +1 for (platelets >=50).

Exclusion Criteria:

1. Has previous treatment for HR MDS or CMML or low-blast AML with chemotherapy or other antineoplastic agents including hypomethylating agent (HMAs) such as decitabine or azacitidine. Previous treatment is permitted with hydroxyurea and with lenalidomide, except that lenalidomide may not be given within 8 weeks before the first dose of study drug.
2. Has acute promyelocytic leukemia as diagnosed by morphologic examination of bone marrow, by fluorescent in situ hybridization or cytogenetics of peripheral blood or bone marrow, or by other accepted analysis.
3. Participants with AML with a WBC count >50,000/mcL. Participants who are cytoreduced with leukapheresis or with hydroxyurea may be enrolled if they meet the eligibility criteria.
4. Is eligible for intensive chemotherapy and/or allogeneic stem cell transplantation. The reason a participant is not eligible for intensive chemotherapy and/or allogeneic stem cell transplantation may consist of one or more of the following factors:

   * Age >75.
   * Comorbidities.
   * Inability to tolerate intensive chemotherapy (e.g., participants with AML with 20%-30% blasts and TRM >=4).
   * Physician decision (e.g., lack of available stem cell donor).
   * The reason a participant is not eligible should be documented in the electronic case report form (eCRF).
5. Has either clinical evidence of or history of central nervous system involvement by AML.
6. Has active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia.
7. Is diagnosed or treated for another malignancy within 2 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease.
8. Has nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection.
9. Has prothrombin time (PT) or aPTT >1.5× upper limit of normal (ULN) or active uncontrolled coagulopathy or bleeding disorder. Participants therapeutically anticoagulated with warfarin, direct thrombin inhibitors, direct factor Xa inhibitors, or heparin are excluded from enrollment.
10. Has known human immunodeficiency virus (HIV) seropositive.
11. Has known hepatitis B surface antigen seropositive, or known or suspected active hepatitis C infection. Note: Participants who have isolated positive hepatitis B core antibody (i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load.
12. Has known hepatic cirrhosis or severe preexisting hepatic impairment.
13. Has known cardiopulmonary disease defined as unstable angina, clinically significant arrhythmia, congestive heart failure (New York Heart Association Class III or IV), and/or myocardial infarction within 6 months before first dose, or severe pulmonary hypertension.
14. Has treatment with strong cytochrome P 3A (CYP3A) inducers within 14 days before the first dose of pevonedistat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (232):
- United States (121):
  - Southern Cancer Center - USOR, Daphne, Alabama
  - Southern Cancer Center - USOR, Mobile, Alabama
  - Southern Cancer Center- USOR, Mobile, Alabama
  - Southeastern Regional Medical Center - CTCA - PPDS, Goodyear, Arizona
  - Arizona Oncology Associates (Orange HOPE) - USOR, Tucson, Arizona
  - Arizona Oncology Associates (Rudasill HOPE) - USOR, Tucson, Arizona
  - Arizona Oncology Associates (Wilmot HOPE) - USOR, Tucson, Arizona
  - Compassionate Care Research Group Inc. at Compassionate Cancer Care Medical Group, Inc, Corona, California
  - Compassionate Cancer Care Medical Group Inc, Fountain Valley, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Emad Ibrahim, MD, Inc, Redlands, California
  - Compassionate Care Research Group Inc. at Compassionate Cancer Care Medical Group, Inc, Riverside, California
  - Rocky Mountain Cancer Centers (Aurora) - USOR, Aurora, Colorado
  - Rocky Mountain Cancer Centers (Boulder) - USOR, Boulder, Colorado
  - Rocky Mountain Cancer Centers (Colorado Springs) - USOR, Colorado Springs, Colorado
  - Quest Diagnostics, INC, Denver, Colorado
  - Colorado Blood Cancer Institute - PPDS, Denver, Colorado
  - Presbyterian Saint Lukes Medical Center Laboratory, Denver, Colorado
  - Presbyterian/St. Luke's Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers (Williams) - USOR, Denver, Colorado
  - Rocky Mountain Cancer Centers (Denver) - USOR, Denver, Colorado
  - Kaiser Foundation Health Plan, Denver, Colorado
  - Laboratory Corporation of America, Englewood, Colorado
  - Rocky Mountain Cancer Centers (Lakewood) - USOR, Lakewood, Colorado
  - Rocky Mountain Cancer Centers (Littleton) - USOR, Littleton, Colorado
  - Rocky Mountain Cancer Centers (Lone Tree) - USOR, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers (Longmont) - USOR, Longmont, Colorado
  - Rocky Mountain Cancer Centers (Parker) - USOR, Parker, Colorado
  - Rocky Mountain Cancer Centers (Pueblo) - USOR, Pueblo, Colorado
  - Rocky Mountain Cancer Centers (Thornton) - USOR, Thornton, Colorado
  - Medstar Research Institute, Washington D.C., District of Columbia
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Altamonte Springs, Florida
  - SCRI Florida Cancer Specialists South, Bonita Springs, Florida
  - SCRI Florida Cancer Specialists South, Bradenton, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Brandon, Florida
  - SCRI Florida Cancer Specialists South, Cape Coral, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Clearwater, Florida
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Gainesville, Florida
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Largo, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Lecanto, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Baptist Health System (N Kendall) - USOR, Miami, Florida
  - SCRI Florida Cancer Specialists South, Naples, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, New Port Richey, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Ocala, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Orange City, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Orlando, Florida
  - SCRI Florida Cancer Specialists South, Port Charlotte, Florida
  - SCRI Florida Cancer Specialists South, Sarasota, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Spring Hill, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, St. Petersburg, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Tampa, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Tavares, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, The Villages, Florida
  - SCRI Florida Cancer Specialists South, Venice, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, Winter Park, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Saint Alphonsus Caldwell Cancer Care Center, Caldwell, Idaho
  - Saint Alphonsus Medical Center, Nampa, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Menorah Medical Center, Overland Park, Kansas
  - Centerpoint Medical Center, Independence, Missouri
  - HCA Midwest Health - SCRI - PPDS, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - New Jersey Hematology Oncology Associates LLC, Brick, New Jersey
  - John Theurer Cancer Center, Hackensack, New Jersey
  - New Jersey Hematology and Oncology, Toms River, New Jersey
  - Weill Cornell Medical Center - Monitoring Location, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Oncology Hematology Care Inc - USOR, Cincinnati, Ohio
  - Fairview Hospital, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oncology Hematology Care, Inc - Fairfield, Fairfield, Ohio
  - Hillcrest Hospital Cancer Care Center, Mayfield, Ohio
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - St. Luke's University Health Network, Easton, Pennsylvania
  - Greenville Health System, Easley, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - Greenville Health System, Greer, South Carolina
  - Greenville Health System, Seneca, South Carolina
  - Greenville Health System, Spartanburg, South Carolina
  - Tennessee Oncology - DICKSON - SCRI - PPDS, Dickson, Tennessee
  - Tennessee Oncology - FRANKLIN - SCRI - PPDS, Franklin, Tennessee
  - Tennessee Oncology - GALLATIN - SCRI - PPDS, Gallatin, Tennessee
  - Tennessee Oncology - SUMMIT - SCRI - PPDS, Hermitage, Tennessee
  - Tennessee Oncology - LEBANON - SCRI - PPDS, Lebanon, Tennessee
  - Tennessee Oncology - MURFREESBORO - SCRI - PPDS, Murfreesboro, Tennessee
  - Sarah Cannon Center for Blood Centers - SCRI - PPDS, Nashville, Tennessee
  - Tennessee Oncolgy - BAPTIST - SCRI - PPDS, Nashville, Tennessee
  - Tennessee Oncology NASH - SCRI - PPDS, Nashville, Tennessee
  - Tennessee Oncology - ST THOMAS WEST - SCRI - PPDS, Nashville, Tennessee
  - Tennessee Oncology SKYLINE - SCRI - PPDS, Nashville, Tennessee
  - Tennessee Oncology - SOUTHERN HILLS - SCRI - PPDS, Nashville, Tennessee
  - Tennessee Oncology - SHELBYVILLE - SCRI - PPDS, Shelbyville, Tennessee
  - Tennessee Oncology - SMYRNA - SCRI - PPDS, Smyrna, Tennessee
  - Texas Oncology (West 38) - USOR, Austin, Texas
  - Texas Oncology (Balcones) - USOR, Austin, Texas
  - Texas Oncology (James Casey) - USOR, Austin, Texas
  - Texas Oncology (Medical City) - USOR, Dallas, Texas
  - Baylor Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology (Tyler) - USOR, Longview, Texas
  - Texas Oncology (E Common) - USOR, New Braunfels, Texas
  - Texas Oncology (Round Rock) - USOR, Round Rock, Texas
  - Texas Oncology - San Antonio Medical Center - USOR, San Antonio, Texas
  - Texas Oncology (Tyler) - USOR, Tyler, Texas
  - Oncology and Hematology Associates of Southwest Virginia (Blacksburg) - USOR, Blacksburg, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Oncology and Hematology Associates of Southwest Virginia (Low Moor) - USOR, Low Moor, Virginia
  - Oncology and Hematology Associates of Southwest Virginia (Roanoke) - USOR, Roanoke, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc, Salem, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Wytheville, Virginia
- Australia (7):
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Icon Cancer Care, South Brisbane, Queensland
  - Icon Cancer Care Southport, Southport, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Liverpool Hospital, Liverpool
- Belgium (5):
  - Algemeen Ziekenhuis Klina, Brasschaat, Antwerpen
  - CHU UCL Namur asbl - Site Godinne, Yvoir, Namur
  - AZ Sint-Jan AV, Bruges, West-Vlaanderen
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Brazil (6):
  - Liga Paranaense de Combate Ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - Liga Norte Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Centro de Pesquisas Oncologicas, Florianópolis, Santa Catarina
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre
  - Universidade Federal do Rio de Janeiro - UFRJ, Rio de Janeiro
  - Hospital Santa Marcelina, São Paulo
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- China (2):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Kralovehradeck Kraj
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- France (4):
  - Hopital Cote de Nacre, Caen, Calvados
  - CHU Angers, Angers, Maine-et-Loire
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Saint Louis, Paris
- Germany (4):
  - Universitatsklinikum Tubingen, Tübingen, Baden-Wurttemberg
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Marien Hospital Akademisches Lehrkrankenhaus, Düsseldorf
- Greece (9):
  - Laiko General Hospital of Athens, Athens, Attica
  - Athens General Hospital 'G Gennimatas', Athens, Attica
  - Attikon University General Hospital, Athens, Attica
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Laiko General Hospital of Athens, Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - University General Hospital of Patras, Pátrai
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Israel (6):
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center PPDS -, Jerusalem
  - Galilee Medical Center, Nahariya
  - ZIV Medical Center, Safed
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Italy (6):
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna, Emilia-Romagna
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia - INCIPIT - PIN, Brescia, Lombardy
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Centro Di Riferimento Oncologico Della Basilicata, Rionero in Vulture
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliero Universitaria San Giovanni Battista Di Torino, Torino
- Japan (15):
  - Japan Mutual Aid Association of Public School Teachers Chugoku Central Hospital, Fukuyama, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Fukushima Medical University Hospital, Fukushima, Hukusima
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Juntendo University Hospital, Bunkyo, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Dokkyo Medical University Hospital, Mibu
  - Nagasaki University Hospital, Nagasaki
  - Osaka Metropolitan University Hospital, Osaka
  - Yokohama City University Hospital, Yokohama
  - University of Fukui Hospital, Yoshida-gun
- Mexico (2):
  - Hematologica Alta Especialidad S.C., Huixquilucan
  - Capital Humano para Investigacion Clinica SC, México
- Poland (7):
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii I Transplantologii, Budynek Centrum Medycyny N, Gdansk, Pomeranian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Zaklad Diagnostyki Obrazowej SOR, Opole
  - Szpital Wojewodzki w Opolu, Opole
  - Swietokrzyskie Centrum Onkologii, Kielce, Świętokrzyskie Voivodeship
- Russia (3):
  - City Clinical Hospital # 40, Moscow
  - Russian Research Institute of Hematology and Blood Transfusion, Saint Petersburg
  - North-West Federal Medical Research Center n.a. V.A. Almazov, Saint Petersburg
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hwasun Hospital, Jeongnam
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (10):
  - ICO lHospitalet Hospital Duran i Reynals, LHospitalet de Llobregat, Barcelona
  - Complejo Asistencial Universitario de Leon, León, Castille and León
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Turkey (Türkiye) (6):
  - Gazi University Medical Faculty Gazi Hospital, Ankara
  - Ege University Medical Faculty, Izmir
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
  - Namik Kemal University, Tekirdağ
  - Karadeniz Technical University Faculty of Medicine, Trabzon
- United Kingdom (4):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Maidstone Hospital, Maidstone, Kent
  - St Bartholomew's Hospital, London
  - Singleton Hospital - PPDS, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ades L, Girshova L, Doronin VA, Diez-Campelo M, Valcarcel D, Kambhampati S, Viniou NA, Woszczyk D, De Paz Arias R, Symeonidis A, Anagnostopoulos A, Munhoz EC, Platzbecker U, Santini V, Fram RJ, Yuan Y, Friedlander S, Faller DV, Sekeres MA. Pevonedistat plus azacitidine vs azacitidine alone in higher-risk MDS/chronic myelomonocytic leukemia or low-blast-percentage AML. Blood Adv. 2022 Sep 13;6(17):5132-5145. doi: 10.1182/bloodadvances.2022007334. PMID 35728048
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b60294db2bf003ab499ea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 130 investigative sites globally from 28 November 2017 to 14 October 2024.
Pre-assignment Details: Participants diagnosed with myelomonocytic, and myelogenous leukemia were randomized into two groups in 1:1 ratio to receive single-agent azacitidine or azacitidine + pevonedistat.
Period: Overall Study
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Started | 227 | 227
Safety Population (Safety Population included all enrolled participants who received at least 1 dose of azacitidine alone or pevonedistat + azacitidine.) | 220 | 223
Completed (Participants were considered to have completed the study if they were followed until death or until the sponsor terminated the study.) | 195 | 199
Not Completed | 32 | 28
Not completed — Withdrawal by Subject | 27 | 17
Not completed — Lost to Follow-up | 2 | 3
Not completed — Reason Not Specified | 3 | 8

BASELINE CHARACTERISTICS:
Population: ITT Population included all participants who were randomized.
Groups:
- Azacitidine 75 mg/m^2: Participants were administered azacitidine 75 mg/m^2 IV or SC injection on Days 1 to 5, Days 8 and 9, in 28-day treatment cycles until disease progression or unacceptable toxicity or up to a maximum of 63 cycles.
- Total: Total of all reporting groups
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 | Total
Number analyzed (Participants) | 227 | 227 | 454
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (8.22) | 73.0 (7.65) | 73 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 95 | 180
  Male | 142 | 132 | 274
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 31 | 57
  Not Hispanic or Latino | 188 | 189 | 377
  Unknown or Not Reported | 13 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 20 | 31 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 189 | 180 | 369
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 10 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 3 | 4 | 7
  Belgium | 8 | 3 | 11
  Brazil | 10 | 18 | 28
  China | 2 | 0 | 2
  Czech Republic | 10 | 6 | 16
  Germany | 6 | 3 | 9
  Spain | 26 | 23 | 49
  France | 13 | 8 | 21
  United Kingdom | 1 | 3 | 4
  Greece | 30 | 28 | 58
  Israel | 6 | 6 | 12
  Italy | 14 | 9 | 23
  Japan | 12 | 26 | 38
  Korea, Republic of | 4 | 2 | 6
  Poland | 11 | 10 | 21
  Russia | 22 | 12 | 34
  Turkey | 5 | 5 | 10
  Canada | 2 | 7 | 9
  Mexico | 2 | 5 | 7
  United States of America | 40 | 49 | 89
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: ITT Population included all participants who were randomized. Number analyzed is the number of participants with data available for height at Baseline.
  centimeter (cm)
    number analyzed (Participants) | 225 | 223 | 448
    (all) | 167.59 (9.439) | 166.31 (10.098) | 166.95 (9.783)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: ITT Population included all participants who were randomized. Number analyzed is the number of participants with data available for weight at Baseline.
  kilogram (kg)
    number analyzed (Participants) | 227 | 226 | 453
    (all) | 77.65 (16.143) | 75.82 (15.996) | 76.73 (16.078)
Body Surface Area [Mean (Standard Deviation); unit: meter square (m^2)] — Body surface area is defined as [height (cm) × weight (kg) / 3600]^1/2 Population: ITT Population included all participants who were randomized. Number analyzed is the number of participants with data available for body surface area at Baseline.
  meter square (m^2)
    number analyzed (Participants) | 225 | 223 | 448
    (all) | 1.89 (0.228) | 1.86 (0.233) | 1.88 (0.231)

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the time from randomization to the date of an EFS event. An EFS event was defined as death or transformation to acute myelogenous leukemia (AML) (World Health Organization [WHO] classification as a participant having greater than 20 % blasts in the blood or marrow and an increase of blast count by 50%), whichever event occurred first, in participants with myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemias (CMML). An EFS event was defined as death in participants with low-blast AML.
Time Frame: From randomization until transformation to acute myeloid leukemia, or death due to any cause: up to approximately 42 months
Population: ITT Population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 227 | 227
months | 15.7 [14.42 to 19.68] | 17.7 [13.63 to 20.24]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; IPSS-R indicates the Revised International Prognostic Scoring System; Test type: Superiority; p = 0.557, Log Rank; P-value comparing EFS between treatment groups was based on the 1-sided Cui-Hung-Wang weighted unstratified log-rank test; Hazard Ratio (HR) = 0.968, 95% CI 2-sided [0.757 to 1.238] — HR:unadjusted stratified Cox proportional hazard regression with stratification(low-blast AML,IPSS-R risk groups=very high,high,or intermediate for HRMDS/CMML),treatment as factor.HR<1:better prevention of EFS in combination arm than azacitidine arm

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to death from any cause.
Time Frame: Up to approximately 6.9 years
Population: ITT Population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 227 | 227
months | 16.8 [14.92 to 20.11] | 20.3 [17.97 to 22.60]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Overall Survival (OS); Test type: Superiority; p = 0.152, Log Rank — P-value comparing OS between treatment groups was based on the 1-sided Cui-Hung-Wang weighted unstratified log-rank test; Hazard Ratio (HR) = 0.888, 95% CI 2-sided [0.709 to 1.113] — HR:unadjusted stratified Cox proportional hazard regression with stratification(low-blast AML,IPSS-R risk groups=very high,high,or intermediate for HRMDS/CMML),treatment as factor.HR<1: longer survival time in combination arm than azacitidine arm

3. Secondary Outcome: Kaplan-Meier Estimates of Six-Month Survival Rate
Description: Kaplan-Meier estimates for the probability (expressed as a percentage) of participants that survived at the end of Month 6 from randomization are presented.
Time Frame: Month 6
Population: ITT Population included all participants who were randomized. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 174 | 174
percentage probability | 0.825 [0.767 to 0.869] | 0.810 [0.752 to 0.856]

4. Secondary Outcome: Kaplan-Meier Estimates of One-Year Survival Rate
Description: Kaplan-Meier estimates for the probability (expressed as a percentage) of participants that survived at the end of the first year from randomization are presented.
Time Frame: Year 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 141 | 137
percentage probability | 0.693 [0.626 to 0.751] | 0.646 [0.578 to 0.706]

5. Secondary Outcome: Thirty-Day Mortality Reported as Number of Participants Who Died Up to Day 30
Description: 30-day mortality was defined as number of participants who died within 30 days from the first dose of study drug.
Time Frame: Up to Day 30
Population: Safety Population included all enrolled participants who received at least 1 dose of azacitidine alone or pevonedistat + azacitidine.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 220 | 223
Participants | 6 | 5

6. Secondary Outcome: Sixty-Day Mortality Reported as Number of Participants Who Died Up to Day 60
Description: 60-day mortality was defined as number of participants who died within 60 days from the first dose of study drug.
Time Frame: Up to Day 60
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 220 | 223
Participants | 15 | 14

7. Secondary Outcome: Time to Acute Myelogenous Leukemia (AML) Transformation in Higher-Risk Myelodysplastic Syndromes (HR MDS), Higher-Risk Chronic Myelomonocytic Leukemias (HR CMML) and HR MDS/CMML Participants
Description: Time to AML transformation in HR MDS and CMML participants was defined as time from randomization to documented AML transformation as determined by the independent review committee (IRC) assessment. Participants who died before progression to AML were censored. Transformation to AML was defined, according to WHO classification, as a participant having 20% blasts in the blood or marrow and increase of blast count by 50%.
Time Frame: From randomization until transformation to AML (up to approximately 42 months)
Population: ITT Population included all participants who were randomized. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis for the given category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 174 | 177
months
  HR MDS Participants: number analyzed (Participants) | 163 | 161
  HR MDS Participants | 35.6 [26.51 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to low number of participants with event. | NA [23.29 to NA] — The median, and upper limit of 95% CI were not estimable due to low number of participants with event.
  HR CMML Participants: number analyzed (Participants) | 11 | 16
  HR CMML Participants | NA [NA to NA] — The median, lower limit, and upper limit of 95% CI were not estimable due to low number of participants with event. | NA [NA to NA] — The median, lower limit, and upper limit of 95% CI were not estimable due to low number of participants with event.
  HR MDS/CMML Participants | 35.6 [29.04 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with event. | NA [24.28 to NA] — The median, and upper limit of 95% CI were not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Time to AML Transformation in HR MDS Participants; Test type: Superiority; p = 0.562, Log Rank — P-value comparing time to AML Transformation between treatment groups was based on 1-sided stratified log-rank test stratified by IPSS-R risk groups of very high, high, or intermediate for HR MDS; Hazard Ratio (HR) = 1.037, 95% CI 2-sided [0.660 to 1.630] — HR:unadjusted stratified Cox proportional HazardRegression with stratification(IPSS-R risk groups=very high,high,or intermediate for HRMDS/CMML),treatment as factor.HR<1:better prevention of AML transformation in combination arm than azacitidine arm
Statistical Analysis 2: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Time to AML Transformation in HR CMML Participants; Test type: Superiority; p = 0.603, Log Rank — P-value comparing time to AML Transformation between treatment groups was based on 1-sided stratified log-rank test stratified by IPSS-R risk groups of very high, high, or intermediate for HR CMML; Hazard Ratio (HR) = 1.512, 95% CI 2-sided [0.068 to 33.773] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Time to AML Transformation in HR MDS/CMML Participants; Test type: Superiority; p = 0.558, Log Rank — P-value comparing time to AML Transformation between treatment groups was based on 1-sided stratified log-rank test stratified by IPSS-R risk groups of very high, high, or intermediate for HR CMML/MDS; Hazard Ratio (HR) = 1.034, 95% CI 2-sided [0.663 to 1.610] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Number of Participants With Complete Remission (CR) and CR+ Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: CR for HR MDS or CMML is defined as <=5% myeloblasts with normal maturation of all cell lines in the bone marrow, and greater than or equal to >=11 gram per deciliter (g/dL) hemoglobin (Hgb),>=100*10^9/liter (/L) platelets (pl),>=1.0*10^9/L neutrophils and 0% blasts in peripheral blood. CR for low-blast AML: morphologic leukemia-free state, neutrophils of more than 1.0*10^9/L and pl of >=100*10^9/L, transfusion independence, and no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery (CRi) for low-blast AML: participants fulfill all of the criteria for CR except for residual neutropenia (<1.0*10^9/L) or thrombocytopenia (pl<100*10^9/L).
Time Frame: From randomization until CR (up to approximately 42 months)
Population: Response-Evaluable Population (REP) included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 206 | 208
Participants | 71 | 63
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Number of Participants With Complete Remission (CR) and CR+Complete Remission with Incomplete Blood Count Recovery (CRi); Test type: Superiority; p = 0.374, Cochran-Mantel-Haenszel — P-value was obtained from a stratified Cochran-Mantel-Haenszel chi-square test stratified by low-blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML; Absolute Rate Difference = -4.18, 95% CI 2-sided [-13.18 to 4.83]

9. Secondary Outcome: Number of Participants With CR and Marrow CR
Description: Disease responses for HR MDS or CMML are based on the International Working Group (IWG) Response Criteria for MDS. CR for HR MDS or CMML is defined as <=5% myeloblasts with normal maturation of all cell lines in the bone marrow, and >=11 g/dL Hgb, >=100*10^9/L platelets (pl), >=1.0*10^9/L neutrophils and 0% blasts in peripheral blood. Marrow CR: Bone marrow: <=5% myeloblasts and decrease by >=50% over pretreatment.
Time Frame: From randomization until CR or marrow CR (up to approximately 42 months)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 206 | 208
Participants | 91 | 87

10. Secondary Outcome: Number of Participants With CR, Partial Remission (PR) and Hematologic Improvement (HI)
Description: Disease responses for HR MDS/CMML based on Modified IWG Response Criteria for MDS. CR: <=5% myeloblasts with normal maturation of all bone marrow cell lines, >=11 g/dL Hgb, >=100*10^9/L pl, >=1.0*10^9/L neutrophils,0% blasts in peripheral blood. Marrow CR: Bone marrow: <=5% myeloblasts and decrease by >=50% over pretreatment. PR: all CR criteria met except bone marrow blasts >=50% decrease over pretreatment but still >5%. HI: Hgb increase >=1.5 g/dL if <11 g/dL; pl increase >=30*10^9/L if baseline>20*10^9/L or increase from <20*10^9/L to >20*10^9/L and by at least 100%; neutrophil increase by 100% and absolute increase of >0.5*10^9/L if baseline <1.0*10^9/L.
Time Frame: From randomization until, CR, PR or HI (up to approximately 42 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 206 | 208
Participants | 77 | 76

11. Secondary Outcome: Number of Participants With CR and Marrow CR and PR
Description: Disease responses for HR MDS/CMML based on Modified IWG Response Criteria for MDS. CR: <=5% myeloblasts with normal maturation of all bone marrow cell lines, >=11 g/dL Hgb, >=100*10^9/L pl, >=1.0*10^9/L neutrophils,0% blasts in peripheral blood. Marrow CR: Bone marrow: <=5% myeloblasts and decrease by >=50% over pretreatment. PR: all CR criteria met except bone marrow blasts >=50% decrease over pretreatment but still >5%.
Time Frame: From randomization until CR or Marrow CR and PR (up to approximately 42 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 206 | 208
Participants | 91 | 87

12. Secondary Outcome: Number of Participants With CR and Marrow CR, PR and Hematologic Improvement (HI)
Description: Disease responses for HR MDS/CMML based on Modified IWG Response Criteria for MDS. CR: <=5% myeloblasts with normal maturation of all bone marrow cell lines, >=11 g/dL Hgb, >=100*10^9/L pl, >=1.0*10^9/L neutrophils,0% blasts in peripheral blood. Marrow CR: Bone marrow: <=5% myeloblasts and decrease by >=50% over pretreatment. PR: all CR criteria met except bone marrow blasts >=50% decrease over pretreatment but still>5%. HI: Hgb increase >=1.5 g/dL if baseline <11 g/dL; pl increase >=30*10^9/L if baseline>20*10^9/L or increases from <20*10^9/L to >20*10^9/L and by at least 100%; neutrophil increases by 100% and absolute increases of >0.5*10^9/L if baseline <1.0*10^9/L.
Time Frame: From randomization until CR, marrow CR, PR or HI (up to approximately 42 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 206 | 208
Participants | 112 | 117

13. Secondary Outcome: Number of Participants With Overall Response (OR)
Description: Disease responses for HR MDS/CMML based on Modified IWG Response Criteria for MDS; for low-blast AML on Revised IWG Response Criteria for AML. Overall response=CR or PR for HR MDS/CMML and CR + CRi + PR for low-blast AML. CR for HR MDS/CMML: <=5% myeloblasts with normal maturation of all bone marrow cell lines, >=11 g/dL Hgb, >=100*10^9/L pl, >=1.0*10^9/L neutrophils, 0% blasts in peripheral blood and PR: all CR criteria met except bone marrow blasts >=50% decrease over pretreatment but still>5%. For low-blast AML-CR:morphologic leukemia-free state>1.0*10^9 neutrophils, >=100*10^9/L pl, transfusion independence, no residual evidence of extramedullary leukemia; CR with incomplete blood count recovery (CRi): fulfill CR criteria except residual neutropenia <1.0*10^9/L or pl <100*10^9/L; PR: all CR hematological values but >=50% decrease in bone marrow aspirate.
Time Frame: From randomization until CR and PR or CR, CRi and PR (up to approximately 42 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 206 | 208
Participants | 73 | 64
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Number of Participants with OR; Test type: Superiority; p = 0.329, Cochran-Mantel-Haenszel — P-value was obtained from a stratified Cochran-Mantel-Haenszel chi-square test stratified by low-blast AML, Revised International Prognostic Scoring System (IPSS-R) risk groups of very high, high, or intermediate for HR MDS/CMML; Absolute Rate Difference = -4.67, 95% CI 2-sided [-13.72 to 4.39]

14. Secondary Outcome: Number of Participants With Overall Response 2 (OR2)
Description: OR2=participant with best overall response of CR+PR+HI in HR MDS/CMML participants,or of CR+CRi+PR in low-blast AML participants.CR:≤5% myeloblasts with normal maturation of all bone marrow(BM)cell lines,≥11g/dL Hgb,≥100*10^9/L pl,≥1.0*10^9/L neutrophils,0% blasts in peripheral blood;PR:all CR criteria met except BM blasts ≥50% decrease over pretreatment but still >5%;HI:Hgb increase(inc) ≥1.5g/dL if baseline(BL)<11 g/dL;pl inc≥30*10^9/L if BL>20*10^9/L or inc from <20*10^9/L to >20*10^9/L and by 100%;neutrophil inc by 100%;absolute inc of >0.5*10^9/L if BL<100*10^9/L.For low-blast AML-CR:morphologic leukemia-free state >1.0*10^9 neutrophils,≥100*10^9/L pl,transfusion independence,no residual evidence of extramedullary leukemia;CR with incomplete blood count recovery:fulfill CR criteria except residual neutropenia <1.0*10^9/L or pl<100*10^9/L;PR:all CR hematological values but ≥50% decrease in BM aspirate.Number of responders determined by independent review committee(IRC) assessment.
Time Frame: From randomization until, CR, PR or HI or CR, CRi or PR (up to approximately 42 months)
Population: REP: all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Data is reported for responders. Three participants were not counted as responders for OR2 as the IRC assessed these participants as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 206 | 208
Participants | 94 | 94
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Number of Participants with OR2; Test type: Superiority; p = 0.891, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]; Absolute Rate Difference = -0.44, 95% CI 2-sided [-10.03 to 9.15]

15. Secondary Outcome: Duration of Complete Remission (CR)
Description: Duration of CR is first documented CR to the first documentation of PD or relapse from CR (participants with low-blast AML) or relapse after CR or PR (participants with HR MDS/CMML). Disease responses for HR MDS or CMML are based on the Modified IWG Response Criteria for MDS and for low-blast AML on the Revised IWG Response Criteria for AML. CR for HR MDS or CMML is defined as <=5% myeloblasts with normal maturation of all cell lines in the bone marrow, and greater than or equal to >=11 g/dL Hgb,>=100*10^9/L pl,>=1.0*10^9/L neutrophils and 0% blasts in peripheral blood. CR for low-blast AML: morphologic leukemia-free state, neutrophils of more than 1.0*10^9/L and pl of >=100*10^9/L, transfusion independence, and no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery (CRi) for low-blast AML: participants fulfill all of the criteria for CR except for residual neutropenia (<1.0*10^9/L) or thrombocytopenia (pl<100*10^9/L).
Time Frame: From CR until first documentation of PD or relapse from CR or relapse after CR or PR (up to approximately 42 months)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Data is reported for participants with complete remission.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 68 | 57
months | 13.1 [6.93 to 29.08] | 17.2 [13.96 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Duration of CR; Test type: Superiority; p = 0.072, Log Rank; P-value was based on 1-sided log-rank test stratified by low-blast AML,IPSS-R risk groups of very high,high,or intermediate for HR MDS/CMML; Hazard Ratio (HR) = 0.679, 95% CI 2-sided [0.402 to 1.146] — Hazard ratio was based on an unadjusted stratified Cox proportional hazard regression model with stratification factors (low-blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML) and treatment as a factor in the model

16. Secondary Outcome: Duration of Complete Remission + Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: Duration of CR is first documented CR to the first documentation of PD or relapse from CR (participants with low-blast AML). Disease responses for low-blast AML were based on the Revised IWG Response Criteria for AML. CR is defined as <=5% myeloblasts with normal maturation of all cell lines in the bone marrow, and greater than or equal to >=11 g/dL hemoglobin (Hgb),>=100*10^9/liter (/L) platelets (pl),>=1.0*10^9/L neutrophils and 0% blasts in peripheral blood. CR for low-blast AML: morphologic leukemia-free state, neutrophils of more than 1.0*10^9/L and pl of >=100*10^9/L, transfusion independence, and no residual evidence of extramedullary leukemia. CR with incomplete blood count recovery (CRi) for low-blast AML: participants fulfill all of the criteria for CR except for residual neutropenia (<1.0*10^9/L) or thrombocytopenia (pl<100*10^9/L).
Time Frame: From CR until first documentation of PD or relapse from CR or relapse after CR or PR (up to approximately 42 months)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Data is reported for participants with CR and CRi.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 15 | 17
months | 8.5 [3.02 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with event. | 15.0 [3.94 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Duration of Complete Remission + Complete Remission with Incomplete Blood Count Recovery (CRi); Test type: Superiority; p = 0.373, Log Rank — P-value comparing duration of CR+CRi between treatment groups was based on 1-sided unstratified log-rank; Hazard Ratio (HR) = 0.846, 95% CI 2-sided [0.306 to 2.339] — Hazard ratio was based on an unadjusted unstratified Cox proportional hazard regression model with treatment as a factor in the model

17. Secondary Outcome: Duration of Overall Response (OR)
Description: Duration of OR: response to first documentation of PD or relapse from CR for low-blast AML or relapse after CR or PR for HR MDS/CMML. Disease responses for HR MDS/CMML based on Modified IWG Response Criteria for MDS; for low-blast AML on Revised IWG Response Criteria for AML. Overall response=CR+PR for HR MDS/CMML and CR+Cri+ PR for low-blast AML.CR for HR MDS/CMML:<=5% myeloblasts with normal maturation of all bone marrow cell lines,>=11 g/dL Hgb,>=100*10^9/L pl,>=1.0*10^9/L neutrophils,0% blasts in peripheral blood and PR:all CR criteria met except bone marrow blasts>=50% decrease over pretreatment but still >5%. For low-blast AML-CR: morphologic leukemia-free state >1.0*10^9 neutrophils,>=100*10^9/L pl, transfusion independence, no residual evidence of extramedullary leukemia; CR with CRi: fulfill CR criteria except residual neutropenia <1.0*10^9/L or pl <100*10^9/L; PR: all CR hematological values but >=50% decrease in % of blasts in bone marrow aspirate.
Time Frame: Up to approximately 42 months
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Data is reported for responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 73 | 64
months | 18.3 [8.31 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with event. | 17.1 [12.68 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Duration of Overall Response (OR); Test type: Superiority; p = 0.320, Log Rank — P-value comparing duration of PR or better response between treatment groups was based on 1-sided log-rank test stratified by low-blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML; Hazard Ratio (HR) = 0.889, 95% CI 2-sided [0.542 to 1.458] — [estimate comment as in outcome 15, analysis 1]

18. Secondary Outcome: Duration of Overall Response 2 (OR2)
Description: Duration of OR2: from date of first documentation of CR+PR+HI to first documentation of PD/relapse after CR/PR for responders of CR+PR+HI for HR MDS/CMML and CR,CRi,PR for low-blast AML. For HR MDS/CMML-CR:<=5% myeloblasts with normal maturation of all bone marrow cell lines,>=11 g/dL Hgb, >=100*10^9/L pl,>=1.0*10^9/L neutrophils, 0% blasts in peripheral blood; PR: all CR criteria met except bone marrow blasts>=50% decrease over pretreatment, still >5%; HI:Hgb inc >=1.5 g/dL if baseline <11 g/dL; pl inc>=30*10^9/L if baseline>20*10^9/L or inc from<20*10^9/L to>20*10^9/L by at least 100%; neutrophil inc by 100% and absolute inc of >0.5*10^9/L if baseline <1.0*10^9/L.For low-blast AML-CR: morphologic leukemia-free state,>1.0*10^9 neutrophils,>=100*10^9/L pl, transfusion independence, no residual evidence of extramedullary leukemia;CRi: fulfill CR criteria except residual neutropenia<1.0*10^9/L or pl <100*10^9/L;PR:all CR hematological values but>=50% decrease in bone marrow aspirate.
Time Frame: Up to approximately 42 months
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 postbaseline disease assessment. Three participants who were non-responders (for OR2) as per the IRC were included in this outcome measure as they had assessment of HI and duration of OR2 for these participants could still be derived based on the pre-specified criteria for HR MDS/CMML participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 95 | 96
months | 18.3 [11.17 to 30.92] | 18.9 [15.01 to NA] — The upper limit of 95% CI was not estimable due to lower number of participants with the event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Duration of Overall Response 2 (OR2); Test type: Superiority; p = 0.151, Log Rank — P-value comparing duration of overall response 2 between treatment groups was based on 1-sided log-rank test stratified by low blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML; Hazard Ratio (HR) = 0.796, 95% CI 2-sided [0.514 to 1.231] — [estimate comment as in outcome 15, analysis 1]

19. Secondary Outcome: Percentage of Participants With Red Blood Cells (RBCs) and Platelet-transfusion Independence
Description: A participant was defined as RBC or platelet-transfusion independent if he/she received no RBC or platelet transfusions for a period of at least 8 weeks before the first dose of study drug through 30 days after the last dose of any study drug. Rate of transfusion independence was defined as number of participants who became transfusion independent divided by the number of participants who were transfusion dependent at Baseline.
Time Frame: Up to approximately 42 months
Population: ITT Population included all participants who were randomized. Overall number analyzed is the number of participants from a subset of the ITT Population who were transfusion dependent at Baseline. Number analyzed is the number of participants who were transfusion dependent at Baseline for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 140 | 129
percentage of participants
  Percentage of Participants With RBCs-transfusion Independence: number analyzed (Participants) | 131 | 122
  Percentage of Participants With RBCs-transfusion Independence | 44.3 | 47.5
  Percentage of Participants With Platelet-transfusion Independence: number analyzed (Participants) | 45 | 33
  Percentage of Participants With Platelet-transfusion Independence | 48.9 | 45.5
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Percentage of Participants With RBC-transfusion Independence; Test type: Superiority; p = 0.573, Cochran-Mantel-Haenszel — P-value was obtained from a stratified Cochran-Mantel-Haenszel chi-square test; Absolute Rate Difference = 3.27, 95% CI 2-sided [-9.02 to 15.55]
Statistical Analysis 2: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Percentage of Participants With Platelet-transfusion Independence; Test type: Superiority; p = 0.477, Cochran-Mantel-Haenszel — P-value was obtained from a stratified Cochran-Mantel-Haenszel chi-square test; Absolute Rate Difference = -3.43, 95% CI 2-sided [-25.84 to 18.97]

20. Secondary Outcome: Duration of Red Blood Cells (RBCs) and Duration of Platelet-transfusion Independence and Duration of Red Blood Cells (RBCs) and Platelet-transfusion Independence
Description: Duration of RBC and platelet transfusion independence was defined as the longest time between the last RBC and/or platelet transfusion before the start of the RBC and/or platelet transfusion-independent period and the first RBC and/or platelet transfusion after the start of the transfusion-independent period, which occurs >= 8 weeks later.
Time Frame: Up to approximately 42 months
Population: ITT Population included all participants who were randomized. Number analyzed is the number of participants who achieved transfusion independence for the specified category, with data available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 227 | 227
months
  Duration of RBC Transfusion Independence: number analyzed (Participants) | 58 | 58
  Duration of RBC Transfusion Independence | 15.6 [10.18 to 28.09] | 13.5 [9.07 to 16.66]
  Duration of Platelet Transfusion Independence: number analyzed (Participants) | 22 | 15
  Duration of Platelet Transfusion Independence | 14.9 [5.09 to 23.23] | 11.6 [2.73 to 16.26]
  Duration of Transfusion Independence: number analyzed (Participants) | 63 | 59
  Duration of Transfusion Independence | 12.0 [8.90 to 19.48] | 13.5 [10.38 to 16.66]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Duration of RBC Transfusion Independence; Test type: Superiority; p = 0.774, Log Rank — P-value comparing duration of RBC or platelet transfusion between treatment groups was based on 1-sided log-rank test stratified by low-blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML; Hazard Ratio (HR) = 1.231, 95% CI 2-sided [0.715 to 2.119] — HR:unadjusted Cox Proportional Hazard regression;stratification(low-blast AML,IPSS-R risk groups=very high,high,intermediate for HRMDS/CMML),treatment as factor.HR<1:longer duration of transfusion independence in combination arm than azacitidine arm
Statistical Analysis 2: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Duration of Platelet Transfusion Independence; Test type: Superiority; p = 0.801, Log Rank — P-value comparing duration of platelet transfusion between treatment groups was based on 1-sided log-rank test stratified by low blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML; Hazard Ratio (HR) = 1.533, 95% CI 2-sided [0.567 to 4.147] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 3: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Duration of Transfusion Independence; Test type: Superiority; p = 0.450, Log Rank — [p-value comment as in outcome 20, analysis 1]; Hazard Ratio (HR) = 0.968, 95% CI 2-sided [0.580 to 1.614] — [estimate comment as in outcome 20, analysis 1]

21. Secondary Outcome: Time to First Complete Remission (CR) or Partial Remission (PR) or Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: Time to first CR or PR is defined as the time from randomization to first documented CR or PR, whichever occurs first. Disease responses for HR MDS or CMML or low-blast AML cycle 6 are based on Modified IWG Response Criteria for MDS and for low-blast AML on Revised IWG Response Criteria for AML. For HR MDS or CMML-CR:<=5% myeloblasts with normal maturation of all bone marrow cell lines,>=11 g/dL Hgb,>=100*10^9/L pl,>=1.0*10^9/L neutrophils, 0% blasts in peripheral blood; PR: all CR criteria met except bone marrow blasts>=50% decrease over pretreatment but still>5%; For low-blast AML-CR: morphologic leukemia-free state,>1.0*10^9/L neutrophils, pl>=100*10^9/L, transfusion independence, no residual evidence of extramedullary leukemia; CR with incomplete blood count recovery: fulfill CR criteria except residual neutropenia<1.0*10^9/L or pl <100*10^9/L; PR: all CR hematological values but with a decrease of at least 50% in the percentage of blasts to 5% to 25% in the bone marrow aspirate.
Time Frame: From randomization until CR or PR (up to approximately 42 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 206 | 208
months | NA [12.12 to NA] — The median, and upper limit of 95% CI was not estimable due to low number of participants with event. | NA [24.61 to NA] — The median, and upper limit of 95% CI was not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Time to First Complete Remission (CR) or Partial Remission (PR) or Complete Remission with Incomplete Blood Count Recovery (CRi); Test type: Superiority; p = 0.228, Log Rank — P-value comparing time to first CR or PR or CRi (low-blast AML) between treatment groups was based on 1-sided stratified log-rank test stratified by low-blast AML,IPSS-R risk groups of very high,high,or intermediate for HR MDS/CMML; Hazard Ratio (HR) = 0.880, 95% CI 2-sided [0.628 to 1.234] — [estimate comment as in outcome 15, analysis 1]

22. Secondary Outcome: Number of Participants With Hematologic Improvement (HI)
Description: Disease responses for HR MDS/CMML based on Modified IWG Response Criteria for MDS. HI: Hgb increase >=1.5 g/dL if baseline <11 g/dL; pl increase >=30*10^9/L if baseline >20*10^9/L or increase from <20*10^9/L to >20*10^9/L by at least 100%; neutrophil increase by 100% and absolute increase of >0.5*10^9/L if baseline <1.0*10^9/L.
Time Frame: From randomization until HI (up to approximately 42 months)
Population: REP included all participants who received at least 1 dose of study drug and had a baseline and at least 1 postbaseline disease assessment. Overall number analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 157 | 163
Participants | 76 | 70
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Number of Participants With HI; Test type: Superiority; p = 0.320, Cochran-Mantel-Haenszel — P-value was obtained from a stratified Cochran-Mantel-Haenszel chi-square test; Absolute Rate Difference = -5.46, 95% CI 2-sided [-16.36 to 5.44]

23. Secondary Outcome: Number of Participants With at Least 1 Inpatient Hospital Admissions Related to HR MDS, CMML or Low-blast AML
Description: Inpatient hospital admission data was collected through transformation to AML (HR MDS/CMML participants) or disease progression (low-blast AML participants) or until initiation of subsequent therapy (all participants), whichever occurred first. Transformation to AML is defined, according to WHO Classification, as a participant having 20% blasts in the blood or marrow and increase of blast count by 50%.
Time Frame: From randomization until transformation to AML or until initiation of subsequent therapy (up to approximately 42 months)
Population: ITT Population included all participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 227 | 227
Participants | 3 | 9
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Number of Participants With at Least 1 Inpatient Hospital Admissions Related to HR MDS, CMML or Low-blast AML; Test type: Superiority; Rate Difference = 2.64, 95% CI 2-sided [-0.30 to 5.58]

24. Secondary Outcome: Time to Progressive Disease (PD), Relapse After CR (Low-blast AML), Relapse After CR or PR (HR MDS/CMML), or Death
Description: Time to PD, relapse after CR(low-blast AML), relapse after CR or PR(HR MDS/CMML), or death,defined as time from date of randomization until date of first documentation of PD,relapse after CR(low-blast AML),relapse after CR or PR(HR MDS/CMML),or death due to any cause, whichever occurs first. In HR MDS/CMML,PD: Participants with<5% blasts:>=50% inc >5% blasts, with 5%-9% blasts:>=50% inc>10% blasts, with 10%-19% blasts:>=50% inc >20% blasts,with 20%-30% blasts, at least 50% decrement from maximum remission/response in granulocytes or pl or reduction in Hgb by>=2 g/dL/new transfusion dependence.Relapse after CR or PR: return to pretreatment bone marrow blast %/Decrement of >=50% from maximum remission/response levels in granulocytes/pl/reduction in Hgb conc.>=1.5 g/dL/transfusion dependence. In AML,PD:>50% inc in bone marrow blasts to >30% blasts,>50% inc in circulating blasts to>30% blasts in peripheral blood, Development of extramedullary disease/new sites of extramedullary leukemia.
Time Frame: From randomization until PD, relapse after CR, or relapse after CR or PR, or death due to any cause, whichever occurs first (up to approximately 42 months)
Population: ITT Population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 227 | 227
months | 11.8 [10.25 to 13.31] | 13.1 [11.01 to 15.84]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Time to Progressive Disease (PD), Relapse after CR (Low-blast AML), Relapse After CR or PR (HR MDS/CMML), or Death; Test type: Superiority; p = 0.084, Log Rank — P-value was obtained from a stratified 1-sided log-rank test stratified by low-blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML; Hazard Ratio (HR) = 0.858, 95% CI 2-sided [0.689 to 1.067] — Hazard ratio was based on a stratified Cox proportional hazard regression model stratified by low-blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML, with treatment as a factor in the model

25. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQOL) Using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire- Core 30
Description: The EORTC QLQ-C30 contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status/QOL scale. Most of the 30 items have 4 response levels (not at all, a little, quite a bit, and very much), with 2 questions relying on a 7-point numeric rating scale. Raw scores are converted into scale scores ranging from 0 to 100. For the functional scales and the global health status/QOL scale, higher scores represent better QOL; for the symptom scales, lower scores represent better QOL. The change from baseline at end of treatment is reported.
Time Frame: Baseline, at approximately 58 months
Population: ITT Population included all participants who were randomized. All participants with PRO measurements at baseline and with data available at end of treatment were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 211 | 210
score on a scale
  Global Health Status/QoL Score: Baseline | 60.3 (22.11) | 61.6 (21.13)
  Global Health Status/QoL Score: Change from Baseline: number analyzed (Participants) | 146 | 124
  Global Health Status/QoL Score: Change from Baseline | -3.0 (25.93) | -8.4 (26.89)
  Physical Functioning Score: Baseline | 69.4 (22.63) | 75.7 (20.38)
  Physical Functioning Score: Change from Baseline: number analyzed (Participants) | 146 | 125
  Physical Functioning Score: Change from Baseline | -7.5 (22.82) | -13.4 (27.51)
  Role Functioning Score: Baseline | 66.9 (30.88) | 73.7 (28.55)
  Role Functioning Score: Change from Baseline: number analyzed (Participants) | 146 | 126
  Role Functioning Score: Change from Baseline | -11.8 (35.41) | -18.3 (36.72)
  Emotional Functioning Score: Baseline | 76.0 (20.96) | 77.6 (22.10)
  Emotional Functioning Score: Change from Baselline: number analyzed (Participants) | 146 | 124
  Emotional Functioning Score: Change from Baselline | -2.5 (23.80) | -5.9 (22.41)
  Cognitive Functioning Score: Baseline | 84.6 (18.29) | 86.1 (17.60)
  Cognitive Functioning Score: Change from Baseline: number analyzed (Participants) | 146 | 125
  Cognitive Functioning Score: Change from Baseline | -7.2 (22.65) | -10.4 (24.38)
  Social Functioning Score: Baseline: number analyzed (Participants) | 211 | 208
  Social Functioning Score: Baseline | 79.3 (25.37) | 78.8 (25.82)
  Social Functioning Score: Change from Baseline: number analyzed (Participants) | 146 | 122
  Social Functioning Score: Change from Baseline | -13.7 (33.89) | -16.5 (34.78)
  Fatigue Score: Baseline | 38.5 (25.44) | 33.8 (24.24)
  Fatigue Score: Change from Baseline: number analyzed (Participants) | 146 | 126
  Fatigue Score: Change from Baseline | 6.6 (26.41) | 12.3 (31.22)
  Nausea/Vomiting Score: Baseline | 4.6 (11.39) | 4.7 (10.96)
  Nausea/Vomiting Score: Change from Baseline: number analyzed (Participants) | 146 | 125
  Nausea/Vomiting Score: Change from Baseline | 2.4 (19.08) | 1.9 (15.00)
  Pain Score: Baseline | 20.9 (25.55) | 19.4 (26.42)
  Pain Score: Change from Baseline: number analyzed (Participants) | 146 | 125
  Pain Score: Change from Baseline | 5.8 (30.36) | 6.8 (33.34)
  Dyspnoea Score: Baseline | 25.4 (29.83) | 24.4 (28.90)
  Dyspnoea Score: Change from Baseline: number analyzed (Participants) | 146 | 124
  Dyspnoea Score: Change from Baseline | 5.9 (28.95) | 5.9 (29.46)
  Insomnia Score: Baseline | 27.2 (27.96) | 25.7 (30.68)
  Insomnia Score: Change from Baseline: number analyzed (Participants) | 145 | 124
  Insomnia Score: Change from Baseline | 3.2 (34.32) | 4.6 (34.09)
  Appetite Loss Score: Baseline | 23.4 (29.29) | 15.6 (23.99)
  Appetite Loss Score: Change from Baseline: number analyzed (Participants) | 146 | 125
  Appetite Loss Score: Change from Baseline | 4.6 (38.68) | 16.0 (34.03)
  Constipation Score: Baseline | 14.7 (24.78) | 13.8 (22.47)
  Constipation Score: Change from Baseline: number analyzed (Participants) | 146 | 125
  Constipation Score: Change from Baseline | 5.5 (29.56) | 5.1 (28.42)
  Diarrhoea Score: Baseline | 7.6 (18.84) | 7.0 (16.75)
  Diarrhoea Score: Change from Baseline: number analyzed (Participants) | 146 | 124
  Diarrhoea Score: Change from Baseline | 3.0 (22.80) | 1.9 (27.65)
  Financial Difficulties Score: Baseline: number analyzed (Participants) | 211 | 208
  Financial Difficulties Score: Baseline | 14.2 (25.37) | 18.4 (26.76)
  Financial Difficulties Score: Change from Baseline: number analyzed (Participants) | 146 | 122
  Financial Difficulties Score: Change from Baseline | 5.9 (27.03) | 7.4 (30.46)
  QLQ-C30 Summary Score: Baseline: number analyzed (Participants) | 211 | 208
  QLQ-C30 Summary Score: Baseline | 77.9 (14.90) | 80.5 (15.08)
  QLQ-C30 Summary Score: Change from Baseline: number analyzed (Participants) | 145 | 120
  QLQ-C30 Summary Score: Change from Baseline | -6.1 (18.84) | -8.6 (17.75)

26. Secondary Outcome: Number of Participants With Overall Response in Participants Who Have TP53 Mutations, 17p Deletions, and/or Are Determined to be in an Adverse Cytogenetic Risk Group
Description: Disease responses for HR MDS/CMML based on Modified IWG Response Criteria for MDS; for low-blast AML on Revised IWG Response Criteria for AML. Overall response=CR + PR for HR MDS/CMML and CR + CRi + PR for low-blast AML. CR for HR MDS/CMML: <=5% myeloblasts with normal maturation of all bone marrow cell lines, >=11 g/dL Hgb, >=100*10^9/L pl, >=1.0*10^9/L neutrophils,0% blasts in peripheral blood and PR: all CR criteria met except bone marrow blasts>=50% decrease over pretreatment but still>5%. For low-blast AML-CR: morphologic leukemia-free state, >1.0*10^9 neutrophils,>=100*10^9/L pl, transfusion independence, no residual evidence of extramedullary leukemia; CR with incomplete blood count recovery (CRi): fulfill CR criteria except residual neutropenia<1.0*10^9/L or pl<100*10^9/L; PR: all CR hematological values but>=50% decrease in the percentage of blasts to 5% to 25% in bone marrow aspirate.
Time Frame: From randomization until CR, CRi and PR (up to approximately 42 months)
Population: ITT Population included all participants who were randomized. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 52 | 54
Participants
  OR: HR MDS/CMML Participants | 14 | 13
  OR: Low-blast AML Participants: number analyzed (Participants) | 37 | 32
  OR: Low-blast AML Participants | 13 | 12
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; OR: HR MDS/CMML Participants; Test type: Superiority; p = 0.683, Cochran-Mantel-Haenszel — P-value for HR MDS/CMML was obtained from a stratified Cochran-Mantel-Haenszel chi-square test; Absolute Rate Difference = -2.85, 95% CI 2-sided [-19.44 to 13.75]
Statistical Analysis 2: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; ORR: Low-blast AML Participants; Test type: Superiority; p = 0.840, Cochran-Mantel-Haenszel — P-value for Low-blast AML was obtained from an unstratified Cochran-Mantel-Haenszel chi-square test; Absolute Rate Difference = 2.36, 95% CI 2-sided [-20.39 to 25.12]

27. Secondary Outcome: Event-Free Survival in Participants Who Have TP53 Mutations, 17p Deletions, and/or Are Determined to be in an Adverse Cytogenetic Risk Group
Description: Event was defined as death or transformation to AML in participants with MDS or CMML, whichever occurred first. Transformation to AML was defined, according to World Health Organization (WHO) Classification as a participant having >20% blasts in the blood or marrow and increase of blast count by 50%. Event was defined as death in participants with low-blast AML.
Time Frame: From randomization until transformation to AML if eligible or death (up to approximately 42 months)
Population: ITT Population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 227 | 227
months | 12.8 [8.44 to 14.32] | 14.6 [9.99 to 18.99]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Event-Free Survival in Participants who have TP53 Mutations, 17p Deletions, and/or are Determined to be in an Adverse Cytogenetic Risk Group; Test type: Superiority; p = 0.240, Log Rank — P-value comparing EFS between treatment groups was based on 1-sided log-rank test stratified by low-blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML; Hazard Ratio (HR) = 0.877, 95% CI 2-sided [0.608 to 1.263] — HR:unadjusted stratified Cox proportional hazard regression with stratification factors (IPSS-R risk groups=very high,high,or intermediate for HRMDS/CMML),treatment as factor.HR<1:better prevention of EFS in combination arm than azacitidine arm

28. Secondary Outcome: Overall Survival in Participants Who Have TP53 Mutations, 17p Deletions, and/or Are Determined to be in an Adverse Cytogenetic Risk Group
Description: OS was calculated from date of randomization to the date of death due to any cause. Participants without documented death at the time of the analysis were censored as of the date the participant was last known to be alive.
Time Frame: From randomization until death (up to approximately 42 months)
Population: ITT Population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 227 | 227
months | 12.8 [10.84 to 14.78] | 16.1 [11.40 to 20.24]
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Overall Survival in Participants who have TP53 Mutations, 17p Deletions, and/or are Determined to be in an Adverse Cytogenetic Risk Group; Test type: Superiority; p = 0.145, Log Rank — P-value comparing OS between treatment groups was based on 1-sided log-rank test stratified by low-blast AML, IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML; Hazard Ratio (HR) = 0.826, 95% CI 2-sided [0.580 to 1.178] — HR:unadjusted stratified Cox proportional hazard regression with stratification factors(IPSS-R risk groups of very high,high,intermediate) and treatment as factor in model.HR<1: longer survival time in combination arm than azacitidine arm

29. Secondary Outcome: Number of Participants With Overall Response by Cycle 6
Description: Responses for HR MDS/CMML are based on Modified International Working Group (IWG) Response Criteria for MDS and for low-blast AML on Revised IWG Response Criteria for AML. Overall response=CR and PR for HR MDS/CMML and CR+CR with incomplete blood count recovery(CRi)+PR for low-blast AML. CR for HR MDS/CMML:<=5% myeloblasts with normal maturation of all bone marrow cell lines,>=11g/dL hemoglobin (Hgb),>=100*10^9/L platelet (pl),>=1.0*10^9/L neutrophils, 0% blasts in peripheral blood, and PR:all CR criteria met except bone marrow blasts >=50% decrease over pretreatment but still >5%. For low-blast AML-CR:morphologic leukemia-free state,>1.0*10^9 neutrophils, >=100*10^9/L pl, transfusion independence, no residual evidence of extramedullary leukemia;CRi:fulfill CR criteria except residual neutropenia <1.0*10^9/L/thrombocytopenia (pl<100*10^9/L); PR:all CR hematological values but>=50% decrease in percentage of blasts to 5%-25% in bone marrow aspirate.
Time Frame: Up to Cycle 6 (up to approximately Day 168)
Population: REP included all participants who received at least 1 dose of study drug and had a Baseline and at least 1 post-baseline disease assessment. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 206 | 208
Participants
  Overall Response for HR MDS/CMML: number analyzed (Participants) | 157 | 163
  Overall Response for HR MDS/CMML | 36 | 29
  Overall Response for Low-blast AML: number analyzed (Participants) | 49 | 45
  Overall Response for Low-blast AML | 13 | 22
Statistical Analysis 1: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Overall Response for HR MDS/CMML; Test type: Superiority; p = 0.261, Cochran-Mantel-Haenszel — P-value was obtained from a stratified Cochran-Mantel-Haenszel chi-square test stratified by IPSS-R risk groups of very high, high, or intermediate for HR MDS/CMML; Absolute Rate Difference = -5.14, 95% CI 2-sided [-13.95 to 3.68]
Statistical Analysis 2: Comparison: Azacitidine 75 mg/m^2 vs Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2; Overall Response for Low-blast AML; Test type: Superiority; p = 0.026, Cochran-Mantel-Haenszel — P-value was obtained from an unstratified Cochran-Mantel-Haenszel chi-square test; Absolute Rate Difference = 22.36, 95% CI 2-sided [3.22 to 41.49]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (up to approximately 6.9 years)
Description: The Safety Population included all participants who received at least 1 dose of study drug (i.e., pevonedistat + azacitidine or single-agent azacitidine).
Arm/Group | Azacitidine 75 mg/m^2 | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2
All-Cause Mortality (participants affected / at risk) | 153/220 | 150/223
Serious Adverse Events (participants affected / at risk) | 145/220 | 156/223
Other Adverse Events (participants affected / at risk) | 207/220 | 210/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine 75 mg/m^2 (N=220) | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 (N=223)
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 10 | 13
Anal abscess (Infections and infestations) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1
C-reactive protein increased (Investigations) | 1 | 0
COVID-19 (Infections and infestations) | 3 | 1
COVID-19 pneumonia (Infections and infestations) | 5 | 1
Cardiac failure (Cardiac disorders) | 2 | 3
Cardiac failure acute (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 6
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 9
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Central nervous system haemorrhage (Nervous system disorders) | 1 | 0
Central nervous system injury (Injury, poisoning and procedural complications) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colonic abscess (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Death (General disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Dementia with Lewy bodies (Nervous system disorders) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Fatigue (General disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 35 | 43
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2
Fungal infection (Infections and infestations) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 3 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hepatic cyst infection (Infections and infestations) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 0
Hyphaema (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Infection (Infections and infestations) | 5 | 1
Influenza (Infections and infestations) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2
Klebsiella bacteraemia (Infections and infestations) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Leukostasis syndrome (Blood and lymphatic system disorders) | 0 | 1
Listeriosis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 6 | 5
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Malaise (General disorders) | 2 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Medical device site inflammation (General disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1
Mucormycosis (Infections and infestations) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 6
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Occult blood (Investigations) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Perichondritis (Infections and infestations) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 25 | 33
Pneumonia aspiration (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Polypoid cystitis (Renal and urinary disorders) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Product contamination microbial (Product Issues) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pure white cell aplasia (Blood and lymphatic system disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 16 | 6
Rectal abscess (Infections and infestations) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory tract infection (Infections and infestations) | 4 | 3
Sepsis (Infections and infestations) | 10 | 6
Septic shock (Infections and infestations) | 6 | 11
Serratia bacteraemia (Infections and infestations) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Sudden death (General disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 3
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 10
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Thrombophlebitis septic (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 7
Viral infection (Infections and infestations) | 1 | 0
Visceral pain (General disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Vulvitis (Infections and infestations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine 75 mg/m^2 (N=220) | Pevonedistat 20 mg/m^2 + Azacitidine 75 mg/m^2 (N=223)
Abdominal pain (Gastrointestinal disorders) | 15 | 22
Abdominal pain upper (Gastrointestinal disorders) | 12 | 13
Abnormal loss of weight (Metabolism and nutrition disorders) | 12 | 7
Alanine aminotransferase increased (Investigations) | 11 | 19
Anaemia (Blood and lymphatic system disorders) | 82 | 78
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 35
Aspartate aminotransferase increased (Investigations) | 11 | 17
Asthenia (General disorders) | 42 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 25
Blood bilirubin increased (Investigations) | 6 | 14
Blood creatinine increased (Investigations) | 14 | 22
Constipation (Gastrointestinal disorders) | 90 | 82
Contusion (Injury, poisoning and procedural complications) | 10 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 39
Decreased appetite (Metabolism and nutrition disorders) | 24 | 38
Diarrhoea (Gastrointestinal disorders) | 51 | 61
Dizziness (Nervous system disorders) | 25 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 22
Fall (Injury, poisoning and procedural complications) | 12 | 13
Fatigue (General disorders) | 33 | 42
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 15
Haemorrhoids (Gastrointestinal disorders) | 6 | 18
Headache (Nervous system disorders) | 20 | 26
Hypertension (Vascular disorders) | 14 | 20
Hyperuricaemia (Metabolism and nutrition disorders) | 15 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 29
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 16
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 17
Hypotension (Vascular disorders) | 12 | 13
Injection site erythema (General disorders) | 20 | 15
Injection site pain (General disorders) | 9 | 12
Insomnia (Psychiatric disorders) | 22 | 21
Leukopenia (Blood and lymphatic system disorders) | 14 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 14
Nausea (Gastrointestinal disorders) | 63 | 78
Neutropenia (Blood and lymphatic system disorders) | 77 | 73
Neutrophil count decreased (Investigations) | 19 | 33
Oedema peripheral (General disorders) | 30 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 18
Platelet count decreased (Investigations) | 22 | 33
Pneumonia (Infections and infestations) | 19 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 15
Pyrexia (General disorders) | 56 | 53
Stomatitis (Gastrointestinal disorders) | 7 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 74 | 71
Upper respiratory tract infection (Infections and infestations) | 21 | 20
Urinary tract infection (Infections and infestations) | 15 | 22
Vomiting (Gastrointestinal disorders) | 46 | 51
White blood cell count decreased (Investigations) | 11 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT03268954/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT03268954/SAP_003.pdf